CLINICAL TRIAL: NCT00056030
Title: A Phase II Study Of Oxaliplatin (OXAL), 5-Fluorouracil (5-FU), Leucovorin (CF), and Cetuximab (C225) For Patients With Unresectable Hepatic Metastases From Metastatic Adenocarcinoma Of The Colon Or Rectum
Brief Title: Combination Chemotherapy Plus Cetuximab in Treating Patients With Liver Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N014A; NCI-2012-02521 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000271923 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cetuximab + oxaliplatin + leucovorin + fluorouracil (Experimental): Patients receive cetuximab IV over 1 hour (over 2 hours on day 1 of course 1 only) on days 1 and 8. Patients also receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-2. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity, for a minimum of 12 courses or until deemed to have resectable disease.
  Quality of life is assessed at baseline and prior to each treatment course.
  Patients are followed every 3 months for 1 year and then every 6 months for 3 years.
  Interventions: Biological: cetuximab; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Biological: cetuximab
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as cetuximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining chemotherapy with cetuximab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with cetuximab works in treating patients with unresectable liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the surgical resectability rate of patients with unresectable hepatic metastases secondary to metastatic colorectal adenocarcinoma treated with oxaliplatin, fluorouracil, leucovorin calcium, and cetuximab.
* Determine the response rate and overall survival of patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 1 hour (over 2 hours on day 1 of course 1 only) on days 1 and 8. Patients also receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-2. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity, for a minimum of 12 courses or until deemed to have resectable disease.

Quality of life is assessed at baseline and prior to each treatment course.

Patients are followed every 3 months for 1 year and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 67-73 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of completely resected primary adenocarcinoma of the colon or rectum

  * No gross or microscopic evidence of residual disease
* Liver metastases, meeting 1 of the following criteria:

  * Not optimally resectable
  * Requires resection of all 3 major hepatic veins, the portal vein bifurcation, or the retrohepatic vena cava
  * Includes the main right or main left portal vein and the main hepatic vein of the opposite lobe
  * Requires more than a right or left trisegmentectomy
  * At least 6 metastatic lesions distributed diffusely in both lobes of the liver
* Measurable disease

  * At least 1 measurable lesion ≥ 20 mm
* No evidence of extrahepatic metastases by physical examination or x-ray
* No previously resected extrahepatic metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ 9 g/dL
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ ULN
* No preexisting chronic hepatic disease (e.g., chronic active hepatitis, cirrhosis) that would preclude surgical resection of metastases

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No myocardial infarction within the past 6 months
* No clinical evidence of congestive heart failure
* No New York Heart Association class III-IV heart disease
* No significant cardiac disease
* No uncontrolled hypertension
* No unstable angina
* No congestive heart failure
* No uncontrolled arrhythmias

Gastrointestinal

* Adequate oral nutrition with estimated caloric intake of ≥ 1,500 calories/day
* No severe anorexia or frequent nausea and/or vomiting
* No history of gastrointestinal bleeding that has not been appropriately addressed

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to tolerate major surgery
* No prior allergic reaction or known sensitivity to chimerized or murine monoclonal antibody therapy
* No documented presence of human anti-mouse antibodies
* No known allergy to other platinum compounds
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer, carcinoma in situ, or tumors associated with less than 10% probability of death within 5 years of diagnosis
* No preexisting neuropathy ≥ grade 2
* No symptomatic pulmonary fibrosis or interstitial pneumonitis
* No uncontrolled bacterial or viral infection
* HIV negative
* No fungal infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No colony-stimulating factors within 24 hours of day 1 of each course
* No concurrent immunotherapy

Chemotherapy

* At least 1 year since prior adjuvant systemic fluorouracil with or without levamisole or with or without leucovorin calcium
* No prior oxaliplatin
* No prior systemic chemotherapy for metastatic disease
* No prior chemoembolization for metastatic disease
* No prior hepatic artery infusion chemotherapy for metastatic disease
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 12 months since prior adjuvant radiotherapy
* Prior radiofrequency ablation allowed
* No prior radiotherapy to the liver
* No prior radiotherapy to more than 25% of the bone marrow
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* More than 21 days since prior abdominal exploration (with or without intestinal resection)

Other

* No prior anti-EGFR-directed therapy
* Prior cryotherapy allowed
* No oral cryotherapy on day 1 of each course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2004-12 (Actual); Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Surgical resectability rate as assessed by surgical resection of liver metastases | Up to 4 years

SECONDARY OUTCOMES:
Response rate as measured by RECIST criteria every 6 weeks | Up to 4 years
Overall survival | Up to 4 years
Quality of life as assessed by UNISCALE and Symptom Distress Scale every 6 weeks | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (162):
- United States (162):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital and Medical Center, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Big Sky Oncology, Great Falls, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin